CLINICAL TRIAL: NCT03007992
Title: Phase II Study of Metronomic Treatment With Daily Oral Vinorelbine as First-line Chemotherapy in Patients With Advanced/Metastatic HR+/HER2- Breast Cancer Resistant to Endocrine Therapy
Brief Title: Metronomic Treatment With Daily Oral Vinorelbine as First-line Chemotherapy in Patients With Advanced/Metastatic Hormone Receptor Positive (HR+)/Human Epidermal Growth Factor Receptor 2 Negative (HER2-) Breast Cancer
Acronym: VinoMetro
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Collaborators: Pierre Fabre Pharma GmbH (Industry)
Responsible Party: Principal Investigator, Marcus Schmidt, MD, Univ.-Prof. Dr. med., Johannes Gutenberg University Mainz
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-007
Record Dates: First submitted 2016-12-15; First posted 2017-01-02 (Estimated); Last update posted 2019-08-12 (Actual); Status verified 2019-02

CONDITIONS: Metastatic Breast Cancer
Keywords: Breast cancer; Vinorelbine; Metronomic chemotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vinorelbine Oral (Experimental): Test product: Navelbine® 20 mg / 30 mg soft capsules
  Interventions: Drug: Vinorelbine

INTERVENTIONS:
Drug: Vinorelbine — Oral vinorelbine will be administered at a daily dose of 30 mg (flat dose without any adaptation to body weight or body surface area) without breaks. Treatment will continue until disease progression, occurrence of unacceptable toxicity, patient's refusal or investigator's decision to stop the treatment.
  Other Names: Navelbine® soft capsules

SUMMARY:
The purpose of the trial is to investigate the efficacy of metronomic treatment with daily oral vinorelbine in terms of clinical benefit rate based on local radiological assessment in patients with advanced/metastatic HR+/HER2- breast cancer resistant to endocrine therapy.

DETAILED DESCRIPTION:
In terms of the chronic nature of advanced/metastatic breast cancer, there is a high medical need for new treatment options after failure of hormonal treatment that prolong the interval to the start of intensive cytotoxic therapy, which is commonly associated with impaired quality of life (QoL) and potentially serious side effects. In this respect, metronomic treatment with daily administration of oral vinorelbine could provide an efficacious treatment option with limited toxicities.

Accordingly, this national, multi-centre, open-label, single-arm phase II trial aims to investigate a truly metronomic schedule with daily oral vinorelbine in HR+/HER2-patients with metastatic breast cancer resistant to endocrine therapy, by assessing efficacy and safety. Oral vinorelbine will be administered at a daily dose of 30 mg (flat dose without any adaptation to body weight or body surface area) without breaks. Treatment will continue until disease progression, occurrence of unacceptable toxicity, patient's refusal or investigator's decision to stop the treatment.

In the course of the study, the following interim and final analyses will be done:

i) 1st interim analysis (safety): This analysis will be performed on the basis of 10 patients, who were initially included into the study and who are eligible for safety evaluation; frequency statistics of (serious) adverse events will be analysed.

ii) 2nd interim analysis (efficacy): This analysis will be performed at the completion of the 1st Simon stage.

iii) Final analysis (complete): This analysis will be performed after completion of the follow-up phase (6 months of follow-up after Last Patient Last Treatment).

ELIGIBILITY:
Inclusion Criteria:

1. Written (personally dated and signed) informed consent prior to the performance of any trial specific procedure
2. Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and/or the follow-up schedule
3. Female patient ≥ 18 years of age
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-1, which the investigator assesses as being stable at time of screening
5. Estimated life expectancy ≥ 16 weeks
6. Histologically confirmed adenocarcinoma of the breast
7. Documented locally advanced or metastatic disease, previously untreated by palliative chemotherapy and not amenable to any curative treatment
8. Hormone receptor positive disease determined by ≥ 1% positive stained cells for oestrogen and/or progesterone receptor by immunohistochemistry on the primary tumour or on a metastatic site
9. HER2-negative disease assessed by 0-1+ immuno-histochemistry (IHC) or 2+ IHC with negative fluorescence in situ hybridization (FISH) or CISH) on the primary tumour or on a metastatic site
10. Availability of archival (from the most recently obtained sample) or fresh tumour tissue from patients included in the trial for the analysis of relevant metronomic biomarkers; one tumour block (preferred) or a minimum of 12 (recommended: 15) unstained slides to be provided
11. Relapse ≤ 12 months from end of adjuvant hormonal therapy or pro¬gres¬sion during/after ≥ 1 line of endocrine therapy in the metastatic set¬ting and/or no longer candidate for further endocrine therapy
12. Prior (neo-)adjuvant chemotherapy is allowed, if the interval between end of chemotherapy and date of registration is > 12 months
13. Prior treatment with everolimus and/or palbociclib in the frame of hormonal therapy is allowed
14. Complete staging before registration (CT/MRI thorax and CT/MRI abdomen/pelvis ≤ 28 days before registration; bone scan ≤ 3 months before registration)
15. Presence of ≥ 1 measurable lesion as per RECIST 1.1, which has not been previously irradiated
16. Adequate bone marrow, hepatic and renal function as defined by the following laboratory values:

    * Absolute neutrophil count (ANC) ≥ 1,500/mm3
    * Platelet count ≥ 100,000/mm3
    * Haemoglobin ≥ 10 g/dL
    * Total serum bilirubin ≤ 1.5 x upper limit of normal (ULN) (≤ 3 x ULN in case of liver metasta¬s¬es)
    * Liver transaminases ≤ 2.5 x ULN (≤ 5 x ULN in case of liver metasta¬s¬es)
    * Alkaline phosphatase ≤ 5 x ULN
    * Creatinine ≤ 1.5 x ULN (creatinine clearance should be assessed based on the Cockcroft-Gault-formula in case of borderline values and should then be ≥ 50 ml/min)
17. Women of childbearing potential must be using a medically accepted method of contraception to avoid pregnancy during 2 months preceding registration, throughout the study period and up to 3 months after last dose of study treatment in such a manner that the risk of pregnancy is minimised; reliable contraception comprises sexual abstinence, male sterilization or double barrier methods (e.g. a combination of male condom with diaphragm).
18. Women of childbearing potential must have a negative serum or urine pregnancy test within 72 hours prior to start of study treatment
19. Ability of the patient to understand the character and the individual consequences of this clinical trial.

Exclusion Criteria:

1. No recovery to ≤ Grade (G)1 side effects (exception: alopecia) of any prior anti-neoplastic treatment
2. Aggressive locally advanced or metastatic breast cancer disease requiring systemic combination therapy
3. Known or suspected central nervous system (CNS) and/or leptomeningeal involvement
4. Current peripheral neuropathy ≥ G2
5. Dysphagia or inability to swallow oral medication
6. Malabsorption syndrome or disease significantly affecting GI-function or major resection of the stomach or proximal small bowel that could affect absorption of oral vinorelbine
7. Other serious illness or medical condition, such as but not limited to:

   * Clinically significant cardiac disease or impaired cardiac function (such as: congestive heart failure requiring treatment (NYHA ≥ II); eft ventricular ejection fraction (LVEF) < 50%; significant cardiac arrhythmia; atrial fibrillation; conduction abnormality such as congenital long QT syndrome or high grade/complete atrioventricular (AV)-blockage; acute coronary syndrome including myocardial infarction, unstable angina pectoris, coronary artery bypass graft, coronary angioplasty or stenting, if < 3 months prior to registration; QTcF > 480 msec at screening)
   * Uncontrolled hypertension (> 140/100 mmHg at rest (average of 3 consecutive readings))
   * Unstable diabetes mellitus
   * Uncontrolled hypercalcemia
   * Clinically significant active infections (current or within the last 2 weeks prior to registration)
   * Previous organ allograft
8. Prior treatment with vinorelbine or other vinca alkaloids
9. Concomitant endocrine therapy (e.g. tamoxifen, aromatase inhibitors, fulvestrant) for advanced breast cancer
10. Concomitant use of yellow-fever vaccination or other attenuated life vaccine
11. Concomitant treatment with strong CYP3A4-inhibitors or strong CYP3A4-inducers (discontinuation before registration is acceptable, if medically feasible and ethically acceptable)
12. Necessity to undergo long-term oxygen therapy
13. Major surgery ≤ 28 days prior to registration and/or no recovery from side effects of such therapy to baseline condition or ≤ G1
14. Radiotherapy ≤ 28 days prior to registration, no recovery from side effects of such therapy to baseline condition or ≤ G1 and/or irradiation of ≥ 30% of bone marrow
15. Known hypersensitivity to vinca alkaloids, soy, peanut or any of the excipients contained in the oral vinorelbine capsules
16. Participation in another clinical trial with any investigational drug ≤ 30 days prior to registration
17. History of another malignancy within the past 5 years prior to registration, except cured basal cell carcinoma of the skin or cured in-situ carcinoma of the cervix
18. Pregnant or nursing (lactating) woman

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-03-02 (Actual); Study Completion 2019-03-02 (Actual)

PRIMARY OUTCOMES:
Clinical Benefit Rate (CBR) | 24 weeks after start of treatment.
  The primary endpoint is the determination of the Clinical Benefit Rate (CBR) at 24 weeks after start of treatment. The response to treatment is measured by computer tomography (CT) or magnetic resonance imaging (MRI) for measurable lesions and evaluation for non-measurable lesions at 24 weeks after start of treatment.

SECONDARY OUTCOMES:
Overall response rate (ORR) | 6 months after last patient last treatment
  Statistical evaluation of above mentioned parameter for each patient measured in duration of month
Disease control rate (DCR) | 6 months after last patient last treatment
  Statistical evaluation of above mentioned parameter for each patient measured in duration of month
Duration of disease control (DoDC) | 6 months after last patient last treatment
  Statistical evaluation of above mentioned parameter for each patient measured in duration of month
Duration of stable disease (DoSD) | 6 months after last patient last treatment
  Statistical evaluation of above mentioned parameter for each patient measured in duration of month
Duration of response (DoR) | 6 months after last patient last treatment
  Statistical evaluation of above mentioned parameter for each patient measured in duration of month
Progression-free survival (PFS) | 6 months after last patient last treatment
  Statistical evaluation of above mentioned parameter for each patient measured in duration of month
Time to treatment failure (TTF) | 6 months after last patient last treatment
  Statistical evaluation of above mentioned parameter for each patient measured in duration of month
Overall survival (OS) | 6 months after last patient last treatment
  Statistical evaluation of above mentioned parameter for each patient measured in duration of month
Number of patients with treatment-related adverse events as assessed by CTCAE v4.0 | 6 months after last patient last treatment
  Determination of frequency and severity of (serious) adverse events and the number of laboratory values worsening from baseline based on the Common Toxicity Criteria (CTC) Grade; other safety data (e.g. vital signs and special tests) will be considered as appropriate
Patient's symptoms and health-related quality of life | 6 months after last patient last treatment
  Evaluation of the Global Health Status/QoL on the basis of the Eastern Cooperative Oncology Group (EORTC) quality of life questionnaire (QLQ)-C30 questionnaire
Histopathological parameters | before start of treatment and upon progression, assessed up to 6 months after last patient last treatment
  Analysis of tumour tissue biomarkers before the start of study treatment and upon progression: histopathological analyses including qualitative assessments of tumor-infiltrating lymphocytes (TIL) involving the evaluation of regulatory T cells (Treg), cluster of differentiation 8 (CD8), CD20 and immune checkpoint parameters (e.g. Programmed Death-Ligand 1 (PD-L1)); additionally, markers like vascular endothelial growth factor-A (VEGF-A), thrombospondin-1 (TSP-1) and hypoxia inducible factor-1 (HIF-1) will be evaluated
Biomarker profiles | before start of treatment, during treatment period and upon progression, assessed up to 6 months after last patient last treatment
  Analysis of blood biomarkers before the start of study treatment, during the treatment period and upon progression: assessment of blood biomarkers, such as CD4+ CD25+ Forkhead-Box-Protein P3 (FOXP3+) Treg, T and B lymphocytes, natural killer (NK) cells and monocytes, hypoxia inducible factor-1 (HIF-1), vascular endothelial growth factor (VEGF), thrombospondin-1 (TSP-1), and to evaluate potential correlations of biomarker expression and clinical outcomes (response, PFS, OS)

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Schmidt, Univ.-Prof. Dr. med., Principal Investigator — Universitätsmedizin Mainz, Klinik und Poliklinik für Geburtshilfe und Frauengesundheit
Locations (8):
- Germany (8):
  - Universitätsklinikum Düsseldorf, Frauenklinik, Düsseldorf
  - Klinikum Frankfurt-Höchst Klinik für Gynäkologie und Geburtshilfe - Operative und konservative Gynäkologie, Gynäkologische Onkologie, Pränataldiagnostik, Geburtshilfe, Frankfurt am Main
  - Universitätsklinikum Halle (Saale), Klinik und Poliklinik für Gynäkologie, Halle
  - Onkologische Schwerpunktpraxis Dr. Karcher, Dr. Fuxius, Dr. Debatin, Heidelberg
  - Universitätsklinikum des Saarlandes, Klinik für Frauenheilkunde, Geburtshilfe und Reproduktionsmedizin, Homburg
  - Universitätsmedizin Mainz, Klinik und Poliklinik für Geburtshilfe und Frauengesundheit, Mainz
  - Klinikum der LMU München, Brustzentrum, München
  - Schwerpunktpraxis für Hämatologie und Onkologie Ravensburg, Ravensburg

REFERENCES:
- [Derived] Krajnak S, Decker T, Schollenberger L, Rose C, Ruckes C, Fehm T, Thomssen C, Harbeck N, Schmidt M. Phase II study of metronomic treatment with daily oral vinorelbine as first-line chemotherapy in patients with advanced/metastatic HR+/HER2- breast cancer resistant to endocrine therapy: VinoMetro-AGO-B-046. J Cancer Res Clin Oncol. 2021 Nov;147(11):3391-3400. doi: 10.1007/s00432-021-03599-2. Epub 2021 Mar 20. PMID 33743073